CLINICAL TRIAL: NCT04563052
Title: Measuring Knowledge and Behavior After an Educational Program on Air Pollution as a Health Risk Reduction Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Villanova University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY-2020-133
Record Dates: First submitted 2020-09-08; First posted 2020-09-24 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Air Pollution, Risk Reduction Behaviors
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education (Experimental): Air pollution educational module exposure.
  Interventions: Behavioral: Educational Program on Air Pollution as a Health Risk Reduction Strategy

INTERVENTIONS:
Behavioral: Educational Program on Air Pollution as a Health Risk Reduction Strategy — A power point presentation about the health impact of exposure to fine particulate matter (PM2.5) on health. Pm2.5 is found outdoors and indoors. Information will be reviewed about steps to take for the participants to locate the information using a smart phone and steps to take to decrease exposure to prevent illness such as heart disease or strokes.

SUMMARY:
Since air pollution contains harmful toxicants, it is important for potential exposure to indoor and outdoor air pollution to be considered as part of an overall health risk reduction strategy. This is a behavioral intervention to assess the effectiveness on an air quality education program in reducing exposure to air pollution and negative health effects. Trial participants will complete a pre-test and home air quality assessment tool. Then, they will participate in an educational module on air quality learn about suggestions to take to avoid exposure and complete a spot test. One month after the educational intervention, the participants will be contacted and asked qualitative questions to assess study effectiveness.

DETAILED DESCRIPTION:
Potential exposure to indoor and outdoor air pollution must be considered as part of an overall health risk reduction strategy. Toxicants identified in outdoor air pollution, fine particulate matter (PM2.5), and photochemical ozone cause a systemic inflammatory response to the heart and lungs after exposure. Inside the home, health issues from exposure to carbon monoxide (CO), PM2.5, nitrogen dioxide (NO2) and volatile organic compounds (VOC) are intensified when the home is sealed with the windows and doors closed. This exploratory study seeks to promote health by teaching participants about strategies to reduce risks related to indoor and outdoor effects of air pollution.

Data collection will consist of an electronic demographic data collection form, home air quality assessment, pre-test and post-test around an educational program and follow-up interview one month after the educational program. Avoidance of air pollution as a health risk reduction method is identified in the literature, however, there is limited research addressing the influence of education on avoidance of environmental toxins as a health risk reduction strategy. Therefore this study will provide a foundation for developing broader educational and behavioral initiatives to improve health outcomes. Due to the COVID-19 pandemic, all aspects of this study will be completed either on-line via the Internet or by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18, speak and read English, have access to a computer or smart phone with Internet access.

Exclusion Criteria:

* Anyone not meeting Inclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Understanding of Educational Intervention | At completion of intervention (one day)
  Participants will be evaluated to determine if they understand the impact of air pollution on health, know how to interpret air quality index information, and how to reduce indoor air pollution.
Implementation of Learned Behaviors During Educational Intervention | One month
  Participants will be assessed for long term understanding of educational intervention and how they have altered their behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Kloster, MSN, RN, Principal Investigator — Villanova University
Locations (1):
- Villanova University, Villanova, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abelsohn A, Stieb DM. Health effects of outdoor air pollution: approach to counseling patients using the Air Quality Health Index. Can Fam Physician. 2011 Aug;57(8):881-7, e280-7. PMID 21841106
- [Background] Brook RD, Franklin B, Cascio W, Hong Y, Howard G, Lipsett M, Luepker R, Mittleman M, Samet J, Smith SC Jr, Tager I; Expert Panel on Population and Prevention Science of the American Heart Association. Air pollution and cardiovascular disease: a statement for healthcare professionals from the Expert Panel on Population and Prevention Science of the American Heart Association. Circulation. 2004 Jun 1;109(21):2655-71. doi: 10.1161/01.CIR.0000128587.30041.C8. PMID 15173049
- [Background] Cascio WE, Davis A, Stone SL. The Green Heart Initiative: using air quality information to reduce adverse health effects in patients with heart and vascular disease. J Cardiovasc Nurs. 2013 Sep-Oct;28(5):401-4. doi: 10.1097/JCN.0b013e318295d1ae. No abstract available. PMID 23938326
- [Background] Chen R, Zhao A, Chen H, Zhao Z, Cai J, Wang C, Yang C, Li H, Xu X, Ha S, Li T, Kan H. Cardiopulmonary benefits of reducing indoor particles of outdoor origin: a randomized, double-blind crossover trial of air purifiers. J Am Coll Cardiol. 2015 Jun 2;65(21):2279-87. doi: 10.1016/j.jacc.2015.03.553. PMID 26022815
- [Background] Di Q, Wang Y, Zanobetti A, Wang Y, Koutrakis P, Choirat C, Dominici F, Schwartz JD. Air Pollution and Mortality in the Medicare Population. N Engl J Med. 2017 Jun 29;376(26):2513-2522. doi: 10.1056/NEJMoa1702747. PMID 28657878
- [Background] Farmer SA, Nelin TD, Falvo MJ, Wold LE. Ambient and household air pollution: complex triggers of disease. Am J Physiol Heart Circ Physiol. 2014 Aug 15;307(4):H467-76. doi: 10.1152/ajpheart.00235.2014. PMID 24929855
- [Background] Laumbach R, Meng Q, Kipen H. What can individuals do to reduce personal health risks from air pollution? J Thorac Dis. 2015 Jan;7(1):96-107. doi: 10.3978/j.issn.2072-1439.2014.12.21. PMID 25694820
- [Background] Ruckerl R, Schneider A, Breitner S, Cyrys J, Peters A. Health effects of particulate air pollution: A review of epidemiological evidence. Inhal Toxicol. 2011 Aug;23(10):555-92. doi: 10.3109/08958378.2011.593587. No abstract available. PMID 21864219
- [Background] Seltenrich N. Take care in the kitchen: avoiding cooking-related pollutants. Environ Health Perspect. 2014 Jun;122(6):A154-9. doi: 10.1289/ehp.122-A154. No abstract available. PMID 24892412
- [Background] Zhang Z, Laden F, Forman JP, Hart JE. Long-Term Exposure to Particulate Matter and Self-Reported Hypertension: A Prospective Analysis in the Nurses' Health Study. Environ Health Perspect. 2016 Sep;124(9):1414-20. doi: 10.1289/EHP163. Epub 2016 May 13. PMID 27177127